CLINICAL TRIAL: NCT02107170
Title: Comparison of Intravenous Anesthetics and Volatile Anesthetics on Postoperative Cognitive Dysfunction of Patients Undergoing Endovascular Repair of Aortic Aneurysm and Endovascular Treatment of Arteriosclerosis Obliterans of Lower Extremities.
Brief Title: Effects of Anesthetics on Postoperative Cognitive Function of Patients Undergoing Endovascular Repair of Aortic Aneurysm and Endovascular Treatment of Arteriosclerosis Obliterans of Lower Extremities.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tao Zhang (Other)
Responsible Party: Sponsor-Investigator, Tao Zhang, Department of anesthesiology, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VIAEV
Record Dates: First submitted 2014-03-25; First posted 2014-04-08 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Endovascular Repair of Aortic Aneurysm; Endovascular Treatment of Arteriosclerosis Obliterans of Lower Extremities
MeSH Terms: interventions — Sevoflurane; Propofol; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Sevoflurane & remifentanil (Experimental): sevoflurane at 0.5 to 1.5 minimum alveolar concentrations plus remifentanil (0.1 - 0.5 µg/kg/min) during the surgery.
  Interventions: Drug: Sevoflurane; Drug: Remifentanil
- propofol & remifentanil (Active Comparator): propofol (50 - 150 µg/kg/min) plus remifentanil (0.1 - 0.5 µg/kg/min) during the surgery.
  Interventions: Drug: Propofol; Drug: Remifentanil

INTERVENTIONS:
Drug: Sevoflurane — sevoflurane-based general anesthesia
  Arms: Sevoflurane & remifentanil
Drug: Propofol — total intravenous anesthesia
  Arms: propofol & remifentanil
Drug: Remifentanil

SUMMARY:
Endovascular repair of aortic aneurysm and endovascular treatment of arteriosclerosis obliterans of lower extremities are two kinds of common surgeries in the investigators' hospital. The effects of anesthetic agents on postoperative outcome, especially cognitive function, are not clear. In this study investigators propose to measure postoperative cognitive function and other outcome of patients who are undergoing these two kinds of surgeries, and try to identify whether there is an association between different kinds of anesthetics and postoperative outcome. Investigators will also observe whether changes in plasma levels of VEGF, TGF-1, TNF-α, IL-1β, and IL-6, are associated with postoperative delirium or cognitive change.

ELIGIBILITY:
Inclusion Criteria:

* age 18-100 years of age
* Patients presenting for Endovascular repair of aortic aneurysm and endovascular treatment of arteriosclerosis obliterans of lower extremities

Exclusion Criteria:

* Patients with pre-existing delirium
* Inablility to converse

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with postoperative cognitive dysfunction | 7 days after surgery

SECONDARY OUTCOMES:
Number of patients with postoperative cognitive dysfunction | 3 months after surgery
Changes in plasma levels of VEGF, TGF-1, TNF-α, IL-1β, and IL-6 (a composite outcome measure) | 3 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China